CLINICAL TRIAL: NCT04454320
Title: Seasonal Variations and Different Treatment Protocols of Intussusception in Children: Our Centers Experiences
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Alaa A.E. Moustafa, MD, Principal Investigator, Minia University
Other Study IDs: intussusception in children
Record Dates: First submitted 2020-06-25; First posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Intussusception
MeSH Terms: conditions — Intussusception

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: INTUSSUSCEPTION IN CHILDREN — the seasonal variation and management outcomes of childhood intussusception.

SUMMARY:
Intussusception remains a common cause of bowel obstruction in children and results in significant morbidity and mortality if not promptly treated. There is a paucity of prospective studies regarding childhood intussusception. This study describes the seasonal variation and management outcomes of childhood intussusception

DETAILED DESCRIPTION:
Intussusception is the invagination of a segment of bowel into an adjacent segment resulting into an intestinal obstruction. It is the most common acquired cause of intestinal obstruction in children aged four months to two years with a peak of incidence between four and nine months of age. Etiology of intussusception is reported to be idiopathic in about 90% of cases and rarely is it associated with pathological lead points such as Meckel's diverticulum, appendix, solid bowel lesions, intestinal polyp, and intestinal lymphoma. It is an occlusive-strangulation type of intestinal obstruction, and all necessary measures should be taken early to ensure prompt diagnosis and treatment to avoid ischaemia and necrosis of bowel. The term comes from two Latin words, intus, which means "inside" and suscipere, which means "to receive". It has been reported in neonates and adults . The ancient Greeks, treated intestinal obstruction with enema or insufflations of air into the anus. Abdominal pain, vomiting and blood in stools are the classic triad and are uncommon and seen in less than one-third of the children affected. Cases often present with non-specific symptoms, including vomiting, pain, irritability, decreased appetite and lethargy, and this may render diagnosis of intussusception difficult. Abdominal ultrasound is considered the standard choice for its diagnosis. Non-surgical management with Pneumatic reduction (PR) by air, hydrostatic reduction by saline or contrast enema is the best procedure.Surgical management by exploratory laparotomy with simple reduction while some cases may require a bowel resection and reanastomosis for gangrenous bowel.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria: The verified diagnosis of intussusceptions in patients by clinical examination and ultrasonography

Exclusion Criteria:

* Patients were excluded if the diagnosis of intussusceptions was not validated or patients who were above 12 years of age.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All pediatric patients (up to 14 years old) hospitalized with diagnosis of bowel intussusception were included in the study.
Sampling Method: Probability Sample
Enrollment: 470 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
the seasonal variation and management outcomes of childhood intussusception. | 2 years
  To evaluate the peak of months recorded to have cases with intussusception in 2 pediatric surgery centers across Egypt To evaluate the different modes of management of intussusception used in our centers.

REFERENCES:
- [Result] Lehnert T, Sorge I, Till H, Rolle U. Intussusception in children--clinical presentation, diagnosis and management. Int J Colorectal Dis. 2009 Oct;24(10):1187-92. doi: 10.1007/s00384-009-0730-2. Epub 2009 May 6. PMID 19418060
- [Result] Parashar UD, Holman RC, Cummings KC, Staggs NW, Curns AT, Zimmerman CM, Kaufman SF, Lewis JE, Vugia DJ, Powell KE, Glass RI. Trends in intussusception-associated hospitalizations and deaths among US infants. Pediatrics. 2000 Dec;106(6):1413-21. doi: 10.1542/peds.106.6.1413. PMID 11099597